CLINICAL TRIAL: NCT05016817
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Idiopathic Pulmonary Fibrosis
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for IPF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-10-ATG-13-08
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; IPF; stem cell treatment
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of Idiopathic pulmonary fibrosis

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe for Idiopathic pulmonary fibrosis (IPF) and can improve the prognosis of afflicted patients. Patients with IPF will receive a single intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease requiring chemotherapeutic drugs such as methotrexate, an autologous T Cell vaccine will be utilized created from the patient's own T cells obtained by apheresis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic Pulmonary Fibrosis
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-03 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: Forced vital capacity (FVC) | Four year follow-up
  It will be completed for each follow up point.
Efficacy: Oxygen saturation test | Four year follow-up
  It will be completed for each follow up point.

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (1):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda

REFERENCES:
- [Background] Averyanov A, Koroleva I, Konoplyannikov M, Revkova V, Lesnyak V, Kalsin V, Danilevskaya O, Nikitin A, Sotnikova A, Kotova S, Baklaushev V. First-in-human high-cumulative-dose stem cell therapy in idiopathic pulmonary fibrosis with rapid lung function decline. Stem Cells Transl Med. 2020 Jan;9(1):6-16. doi: 10.1002/sctm.19-0037. Epub 2019 Oct 15. PMID 31613055
- [Background] Fishman JE, Kim GJ, Kyeong NY, Goldin JG, Glassberg MK. Intravenous stem cell dose and changes in quantitative lung fibrosis and DLCO in the AETHER trial: a pilot study. Eur Rev Med Pharmacol Sci. 2019 Sep;23(17):7568-7572. doi: 10.26355/eurrev_201909_18877. PMID 31539148